CLINICAL TRIAL: NCT00466609
Title: Pharmacological Augmentation Strategies for Obsessive Compulsive Disorder Patients Non-respondent to First Line Medication Treatment: a Double Blind Placebo Controlled Study
Brief Title: Using Drug Augmentation to Treat Obsessive Compulsive Disorder Patients Who Did Not Respond to Previous Treatment
Acronym: EPMTOC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Novartis (Industry)
Responsible Party: Principal Investigator, Juliana Belo Diniz, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05/55628-8; 2005/55628-08 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Obsessive Compulsive Disorder
Keywords: clomipramine; quetiapine; fluoxetine; placebo; augmentation; obsessive compulsive disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Clomipramine; Fluoxetine; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Quetiapine (fluoxetine plus quetiapine) (Experimental): fluoxetine up to 40mg once a day plus Quetiapine up to 200mg once a day, during 12 weeks
  Interventions: Drug: Quetiapine (fluoxetine plus quetiapine)
- Clomipramine (fluoxetine plus clomipramine) (Active Comparator): Fluoxetine up to 40mg once a day plus clomipramine up to 75mg once a day, during 12 weeks
  Interventions: Drug: Clomipramine (fluoxetine plus clomipramine)
- Placebo (fluoxetine plus placebo) (Placebo Comparator): Fluoxetine up to 80 mg once a day plus placebo 3 pills once a day, during 12 weeks
  Interventions: Drug: Placebo (fluoxetine plus placebo)

INTERVENTIONS:
Drug: Clomipramine (fluoxetine plus clomipramine) — Clomipramine at maximum dosage of 75mg per day plus fluoxetine at maximum dosage of 40mg per day
  Other Names: Anafranil
  Arms: Clomipramine (fluoxetine plus clomipramine)
Drug: Quetiapine (fluoxetine plus quetiapine) — Quetiapine at maximum tolerated dosage of 200mg per day plus fluoxetine at maximum dosage of 40mg per day
  Other Names: Seroquel
  Arms: Quetiapine (fluoxetine plus quetiapine)
Drug: Placebo (fluoxetine plus placebo) — Placebo plus fluoxetine at maximum dosage of 80mg per day
  Other Names: Prozac; Daforin (EMS pharmaceutics)
  Arms: Placebo (fluoxetine plus placebo)

SUMMARY:
This will be a controlled, randomized, double-blind and double-dummy study on the treatment augmentation strategy for obsessive compulsive disorder patients non-respondent to first line pharmacological treatment. The investigators will compare: fluoxetine maintenance at maximum dosage for additional 12 weeks; the association of fluoxetine with quetiapine; and the association of fluoxetine with clomipramine.

DETAILED DESCRIPTION:
Arm 1: SSRI (Fluoxetine 40mg* once a day) + Clomipramine 75mg* once a day.

Arm 2: SSRI (Fluoxetine 40mg* once a day) + Quetiapine 200mg* once a day.

Arm 3: SSRI (Fluoxetine 80mg* once a day) + Placebo once a day.

*or maximum tolerated dose

We hypothesize that quetiapine and clomipramine will be effective augmentation strategies for resistant OCD patients in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. OCD diagnosis
2. YBOCS score ≥ 16 (for patients with both obsessions and compulsions) or ≥ 10 (for patients with only obsessions or compulsions)
3. Previously signed informed consent to participate in this clinical trial

Exclusion Criteria:

1. Patients with clinical or neurological diseases that may be worsen by the medications included in treatment protocol
2. Current substance dependence or abuse
3. Current psychotic symptoms
4. Current suicide risk
5. Current pregnancy or intention to get pregnant before the end of the treatment protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
YBOCS | 12 weeks
  Rates of improvement after 12 weeks of treatment based on the difference of initial and final Yale Brown Obsessive Compulsive Scale (YBOCS) scores for obsessions and compulsions

SECONDARY OUTCOMES:
QoL | 12 weeks
  Improvement of quality of life (QOL) will be assessed through SF-36 administered on weeks 0 and 12.
Social Adaptation | 12 weeks
  Improvement of social adaptation using the Social Adaptation Scale (SAS) (Weissman & Payket, 1974) administered on weeks 0 and 12
Tolerability | weeks 0,1,2,3,4,8,12
  Tolerability of the proposed treatments through adverse events follow-up performed each visit (emphasis in serotonergic syndrome)
BDI | 12 weeks
  Score obtained with Beck depression inventory (BDI)
BAI | 12 weeks
  Score obtained with Beck´s anxiety inventory (BAI)
CGI | 12 weeks
  Clinical global impression measure of improvement
Cardiotoxicity | 2 weeks
  Change from baseline EKG regarding QT interval
Plasma levels | weeks 2 and 12
  Fluoxetine dosage and Clomipramine plasmatic dosages (when applies)

CONTACTS AND LOCATIONS:
Overall Officials: Juliana B Diniz, MD, Principal Investigator — University of Sao Paulo Medical School
Locations (1):
- Institute of Psychiatry, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Diniz JB, Shavitt RG, Fossaluza V, Koran L, Pereira CA, Miguel EC. A double-blind, randomized, controlled trial of fluoxetine plus quetiapine or clomipramine versus fluoxetine plus placebo for obsessive-compulsive disorder. J Clin Psychopharmacol. 2011 Dec;31(6):763-8. doi: 10.1097/JCP.0b013e3182367aee. PMID 22020357
- [Derived] Fossaluza V, Diniz JB, Pereira Bde B, Miguel EC, Pereira CA. Sequential allocation to balance prognostic factors in a psychiatric clinical trial. Clinics (Sao Paulo). 2009;64(6):511-8. doi: 10.1590/s1807-59322009000600005. PMID 19578654
- See also: Institutional site of main sponsor — http://www.ipqhc.org.br/
- See also: Main results — https://www.ncbi.nlm.nih.gov/pubmed/22020357
- See also: Secondary analysis results — https://www.ncbi.nlm.nih.gov/pubmed/24288238